CLINICAL TRIAL: NCT00680147
Title: HPV Vaccination Acceptance by African-American Parents: Identifying Psychosocial Barriers
Brief Title: Human Papillomavirus (HPV) Vaccination Acceptance by African-American Parents: Identifying Psychosocial Barriers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Principal Investigator, Peter A. Vanable, Professor, Syracuse University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IISP ID# 33546
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: HPV
Keywords: HPV; Gardasil; African-American; adolescent; health behavior; sexually transmitted infections; This will enroll 300 mothers of teenage girls and boys to identify barriers to HPV vaccination among low-income, African-American teens.
MeSH Terms: conditions — Health Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief HPV vaccine informational intervention (Experimental): Because we anticipated that knowledge and awareness of the HPV vaccine would be low in our study population, our CASI survey included a brief, informational overview of key facts concerning HPV vaccination prior to assessing vaccine acceptance, perceived barriers to vaccination, and intentions to vaccinate. The overview lasted approximately 3 minutes and consisted of a brief overview of key HPV vaccination facts that were presented visually (on the computer screen) and read aloud using a digital recording. HPV and vaccine knowledge, awareness, and attitudes items were administered prior to participants hearing the informational overview.
  Interventions: Behavioral: brief informational intervention to promote HPV vaccine acceptance

INTERVENTIONS:
Behavioral: brief informational intervention to promote HPV vaccine acceptance — Teen and parent participants will receive a brief informational intervention that provides basic facts about the HPV vaccine, including the health benefits and three-dose requirements, along with information regarding where to go to receive the vaccination. A coupon for a free HPV vaccination will provided to the parent for use by their teenage daughter.

SUMMARY:
This will enroll 300 mothers of teenage girls and boys to identify barriers to HPV vaccination among low-income, African-American teens.

DETAILED DESCRIPTION:
The HPV vaccine offers hope that the incidence of cervical cancer can be greatly reduced in the U.S. and globally. However, because the vaccine is recommended for children and early adolescents, vaccine awareness and acceptance among parents is critical to insuring vaccine uptake and public health benefit. Although culturally specific concerns may reduce HPV vaccination among African-American youth, research has not addressed this possibility. Accordingly, the proposed study will enroll 300 mothers in a study to identify barriers to HPV vaccination among low-income, African-American teens. Surveys assessing culturally-specific barriers to HPV vaccination acceptance will be administered to both parents and their vaccine-eligible children. Upon completion of the survey, parents with vaccine-eligible daughters will be invited to receive a free HPV vaccination for their child through a local, teen-friendly health clinic. Outcome analyses will focus on identification of predictors of completed vaccinations among girls and barriers to vaccine acceptance among mothers of teenage sons. Our study will provide critically important behavioral outcome data linking barriers to vaccination to subsequent vaccination decisions in a real-world, health care setting.

ELIGIBILITY:
Inclusion Criteria:

* Females parent or guardian with an African-American daughter or son between the ages of 11 and 17
* African-American adolescents between the ages of 11-17

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2008-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
completed vaccination with Gardasil | 6 months

SECONDARY OUTCOMES:
assessed cross-sectionally, at time of initial enrollment | assessed at time of baseline assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health and Behavior, Syracuse University, Syracuse, New York, United States